CLINICAL TRIAL: NCT05376085
Title: An Open-Label, Randomized, Fasting Condition, Single-dose, Cross-over Study to Evaluate the Bioequivalence "DA-5215 Tab" and "DA-5215-R Tab" in Healthy Volunteers
Brief Title: Bioequivalence Study Between "DA-5215 Tab" and "DA-5215-R Tab"
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DTC21-IP064
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Crossover Assignment single-dose, 2-sequence, 2-period Bioequivalence Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT (Experimental): T: "DA-5215" R: "DA-5215-R"
  Interventions: Drug: DA-5215 Tab; Drug: DA-5215-R Tab
- TR (Experimental): T: "DA-5215" R: "DA-5215-R"
  Interventions: Drug: DA-5215 Tab; Drug: DA-5215-R Tab

INTERVENTIONS:
Drug: DA-5215 Tab — single oral administration of 1 tablet of "DA-5215 Tab" with 150mL water
Drug: DA-5215-R Tab — single oral administration of 1 tablet of "DA-5215-R Tab" with 150mL water

SUMMARY:
An Open-Label, Randomized, Fasting Condition, Single-dose, Cross-over Study to Evaluate the Bioequivalence between "DA-5215 Tab" and "DA-5215-R Tab" in Healthy Volunteers

DETAILED DESCRIPTION:
1. Study design: An open-Label, randomized, 2-sequence, 2-period, fasting condition, single-dose, per oral, cross-over study
2. Administration method:

   The subject should maintain a minimum of 10 hours of fasting status before administration, and give an oral dose of 1 tablet (DA-5215 or DA-5215-R) with 150 mL of water at around 8 a.m. on 1D of each period. The subject should not chew or break the drug, but should swallow in whole with water. The difference in administration time between the subjects is about one minute apart, considering the blood collection time.
3. Wash out period: at least 7 days
4. Blood collection time: Before the administration,15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48 hours after the administration (total 16 times)

ELIGIBILITY:
Inclusion Criteria:

1. A person who aged 19 or older at the time of screening
2. BMI of 18 to 30 (BMI calculation: kg/m2)

   - Males weighing 50kg or more, Females weighing 45kg or more
3. No congenital or chronic diseases or pathological symptoms
4. A person who is judged to be suitable for the study by the investigator based on the clinical laboratory examination
5. A person who agreed to use contraception from the first administration of IP to a week after the last administration of IP
6. A person who has fully understood the contents of the consent form for the study and signed the consent form voluntarily and recorded the date of signature

Exclusion Criteria:

1. A person who has taken a drug that significantly induces (e.g., barbital) or inhibits the drug metabolic enzyme within 30 days prior to the first administration of IP
2. A person who has participated in other clinical trials within six months prior to the first administration of the IP
3. A person who has had whole blood transfusion within 8 weeks or the apheresis within 2 weeks before the first administration of IP
4. A person who has medical history of gastric resection that can affect the drug absorption
5. A person with a history of regular alcohol intake within a month prior to the first administration of the IP:

   * Male: More than 21 cups/week
   * Female: More than 14 cups/week (1 cup: 50 ml of soju, 250 ml of beer, 30ml of spirits)
6. A person who is hypersensitive to any of the IP components
7. A person who has medical history of mental disease
8. A person who is judged not to be suitable for the study by the investigator
9. Lactating or possibly pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Area Under the plasma Concentration versus time curve(AUCt) | Pre-dose ~ 48hours
  Area Under the plasma Concentration versus time curve(AUCt)
Peak Plasma Concentration(Cmax) | Pre-dose ~ 48hours
  Peak Plasma Concentration(Cmax)

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity(AUC∞) | Pre-dose ~ 48hours
  Area under the plasma drug concentration-time curve from time 0 to infinity(AUC∞)
Terminal phase of Half-life(t1/2) | Pre-dose ~ 48hours
  Terminal phase of Half-life(t1/2)
Time of peak concentration(Tmax) | Pre-dose ~ 48hours
  Time of peak concentration(Tmax)
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity(AUCt/AUC∞) | Pre-dose ~ 48hours
  Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity(AUCt/AUC∞)

CONTACTS AND LOCATIONS:
Overall Officials: SeungHyun Kang, Ph.D, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea